CLINICAL TRIAL: NCT04184869
Title: A Multi-Center, Open-Label, Extension Study to Allow Continued Treatment of Patients Who Have Participated in Spectrum-Sponsored Clinical Studies With Belinostat
Brief Title: Extension Study for Patients Who Had Not Met Criteria for Discontinuation in Previous Sponsored Belinostat Trials
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Collaborators: Axis Clinicals Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPI-BEL-502
Record Dates: First submitted 2019-02-07; First posted 2019-12-04 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Solid Tumor; Hematological Malignancies
Keywords: Belinostat; beleodaq; Belinostat treatment extension
MeSH Terms: conditions — Hematologic Neoplasms | interventions — belinostat; Atazanavir Sulfate

STUDY DESIGN:
Intervention Model Description: An extension Study for Patients Who Had Not Met Criteria for Discontinuation in Previous Sponsored Belinostat Trials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Wild Type UGT1A1 (Other): Cohort A: Wild Type, UGT1A1, Belinostat IV Dose: 1000 mg/m2 Frequency: 30-minute infusion once daily from Day 1 to Day 5 of a 21-day cycle.
  Duration: Up to five 21-day cycles (15 weeks) Treatment Period: Up to a total of six 21-day cycles (18 weeks) of treatment total from both the original study protocol and this extension protocol.
  Interventions: Drug: Belinostat
- Heterozygous UGT1A1*28 (Other): Cohort B: Heterozygous, UGT1A1, Belinostat IV Dose: 1000 mg/m2 Frequency: 30-minute infusion once daily from Day 1 to Day 5 of a 21-day cycle.
  Duration: Up to five 21-day cycles (15 weeks) Treatment Period: Up to a total of six 21-day cycles (18 weeks) of treatment total from both the original study protocol and this extension protocol.
  Interventions: Drug: Belinostat
- Homozygous UGT1A1*28 (Other): Cohort C: Homozygous, UGT1A1, Belinostat IV Dose: 750 mg/m2 Frequency: 30-minute infusion once daily from Day 1 to Day 5 of a 21-day cycle.
  Duration: Up to five 21-day cycles (15 weeks) Treatment Period: Up to a total of six 21-day cycles (18 weeks) of treatment total from both the original study protocol and this extension protocol.
  Interventions: Drug: Belinostat
- Belinostat & Atazanavir (Other): Arm: Homozygous UGT1A1*28 genotype subjects with Belinostat IV & Atazanavir
  Dose: 750mg/ m2 (Belinostat IV), 400mg (Atazanavir)
  Frequency: two cycles of 21 days (Belinostat administered through Cycle 2, Day 5) Atazanavir 400mg administered Cycle 1 Day 15 to Day 21, and Cycle 2 Day 1 to Day 5
  Duration: Up to five 21-day cycles (15 weeks) Treatment Period: Up to a total of six 21-day cycles (18 weeks) of treatment total from both the original study protocol and this extension protocol.
  Interventions: Drug: Belinostat; Drug: Atazanavir

INTERVENTIONS:
Drug: Belinostat — Patients can continue to receive belinostat treatment as described in the original study protocol or can be treated per the Investigator's standard of care.
  Belinostat Dose Cohort A & B: 1000mg/m2 Belinostat Dose Cohort C: 750mg/m2 Frequency: once cycle of 21 days: cycle 1, Day 1 and Cycle1, Day 2 to Day 5
  Dose modifications to belinostat during treatment on this extension protocol will be in accordance with the belinostat package insert.
  All patients who receive at least one dose of belinostat treatment in this extension study will be followed for safety through 35 (+/-5) days after their last dose of the treatment or until all treatment related AEs have resolved or returned to Baseline/Grade I, whichever is longer, or until it is determined by the treating physician that the outcome will not change with further follow-up.
  Other Names: beleodaq
Drug: Atazanavir — Patients can continue to receive belinostat treatment as described in the original study protocol or can be treated per the Investigator's standard of care.
  Dose: 750mg/ m2 (Belinostat IV), 400mg (Atazanavir) Frequency: two cycles of 21 days (Belinostat administered through Cycle 2, Day 5) Atazanavir 400mg administered Cycle 1 Day 15 to Day 21, and Cycle 2 Day 1 to Day 5
  Dose modifications to belinostat during treatment on this extension protocol will be in accordance with the belinostat package insert.
  All patients who receive at least one dose of belinostat treatment in this extension study will be followed for safety through 35 (+/-5) days after their last dose of the treatment or until all treatment related AEs have resolved or returned to Baseline/Grade I, whichever is longer, or until it is determined by the treating physician that the outcome will not change with further follow-up.
  Other Names: Reyataz
  Arms: Belinostat & Atazanavir

SUMMARY:
This is an open-label, extension protocol designed to allow patients to continue to receive belinostat treatment after they have completed the protocol-specified assessments and procedures in a Spectrum sponsored belinostat study and have not met the criteria for treatment discontinuation in those studies. This extension of belinostat treatment allowance is not a part of the primary efficacy assessments for those trials. The extension is intended to provide all possible benefits to patients who are having a positive response to belinostat and must be under the Investigator's care. The additional treatment is optional and voluntary.

DETAILED DESCRIPTION:
This is an open-label, extension protocol designed to allow patients to continue to receive belinostat treatment after they have completed the protocol-specified assessments and procedures in a Spectrum sponsored belinostat study and have not met the criteria for treatment discontinuation in those studies. This extension of belinostat treatment allowance is not a part of the primary efficacy assessments for those trials. The extension is intended to provide all possible benefits to patients who are having a positive response to belinostat and must be under the Investigator's care. The additional treatment is optional and voluntary.

This protocol will be available for all patients who have completed the protocol-specified assessments and procedures in Spectrum sponsored belinostat studies. Patients can receive belinostat treatment according to the treatment schedule that is being administered at the time they complete participation in the original clinical study protocol or can be treated per the Investigator's standard of care. Doe modifications during treatment on this extension protocol will be in accordance with the U.S. package insert.

Safety will continue to be followed during the extended belinostat treatment. Therapeutic benefits or efficacy will be followed to the extent that is evaluated according to the institution's standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patient has participated in, and completed, a Spectrum-sponsored clinical study with belinostat and did not meet the treatment discontinuation criteria in the study
* Investigator considers this extended belinostat treatment is appropriate for patient, and patient is suitable for the treatment
* Patient agrees to continue belinostat treatment as defined in the original clinical study protocol
* Patient must be willing to give written Informed Consent and must be able to adhere to dosing and visit schedules and meet study requirements
* Patient is willing to practice two forms of contraception, one of which must be a barrier method, from study entry until at least 30 days after the last dose of the study drug

Exclusion Criteria:

* Patient has an active uncontrolled infection, underlying medical condition, or other serious illness that would impair the ability of the patient to receive belinostat benefit
* Patient is receiving any other treatment modalities including investigational products for their malignancy
* Patient has any medical or non-medical condition that may not be suitable for belinostat treatment, as determined by the investigator and according to the US package insert
* Patient is pregnant or is breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety include assessment of all SAEs, and all deaths on study or within 35 (±5) days of last study treatment | 35 (±5) days after the last dose of belinostat
  Frequency of adverse events (AEs & serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Erard Gilles, MD, Study Director — Navitas Life Sciences Inc.
Locations (1):
- John Wayne Cancer Institute @ Providence Saint John's Health Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No